CLINICAL TRIAL: NCT05283512
Title: Intravenous vs. Oral Hydration to Reduce the Risk of Post-Contrast Acute Kidney Injury After Intravenous Contrast-Enhanced Computed Tomography in Patients With Severe Chronic Kidney Disease (ENRICH): A Randomized Controlled Trial
Brief Title: Intravenous vs. Oral Hydration to Reduce the Risk of Post-Contrast Acute Kidney Injury After Intravenous Contrast-Enhanced Computed Tomography in Patients With Severe Chronic Kidney Disease
Acronym: ENRICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Department of Nephrology, Odense University Hospital (Unknown); Department of Clinical Genetics, Odense University Hospital (Unknown); The A.P. Moller Foundation (Unknown); The Research Counsil of Odense University Hospital (Unknown); Copenhagen University's Research Foundation for Medical Students (Unknown); Helen and Ejnar Bjørnow's Foundation (Unknown); Novo Nordisk A/S (Industry); Sophus Jacobsen and Astrid Jacobsen's Foundation (Unknown); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Emil Johannes Ravn, Medical student and clinical research assistant, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-20210126; Danish Data Protection Act (Registry Identifier: 21/66779)
Record Dates: First submitted 2022-02-25; First posted 2022-03-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-03

CONDITIONS: Contrast-induced Nephropathy; Kidney Injury; Kidney Failure, Chronic; Risk Reduction
Keywords: Intravenous; Contrast material; Computed Tomography; Cardiac CT; Prophylaxis; Oral Hydration; IV-hydration
MeSH Terms: conditions — Kidney Failure, Chronic; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Patients are allocated to either oral- or IV-hydration
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV-hydration group (standard of care according to international guidelines) (Other): The IV-hydration with isotonic 0.9% NaCl will be initiated three hours prior to the IV CECT and completed four hours after IV CECT (infusion rate of 1-3 mL/kg/hour). Patients are prescribed a fixed volume of 1000 mL, which is equally distributed before and after IV CECT (500 mL before and 500 mL after).
  Patients with heart failure (LVEF ≤ 40%) are prescribed a reduced volume of 500 mL, which is also equally distributed before and after IV CECT (250 mL before and 250 mL after).
  Interventions: Other: Preventive treatment with IV-hydration
- Oral hydration group (Active Comparator): The oral hydration regimen will be initiated one-two hours prior to IV CECT and completed within four hours after IV CECT. Patients are prescribed a fixed volume of 1000 mL, which is distributed equally before and after IV CECT (500 mL before and 500 mL after).
  Patients with heart failure (LVEF ≤ 40%) are prescribed a reduced volume of 500 mL, which is equally distributed before and after IV CECT (250 mL before and 250 mL after).
  Interventions: Other: Preventive treatment with oral hydration

INTERVENTIONS:
Other: Preventive treatment with IV-hydration — IV hydration with isotonic 0.9% NaCl
  Arms: IV-hydration group (standard of care according to international guidelines)
Other: Preventive treatment with oral hydration — Oral hydration with regular bottled water
  Arms: Oral hydration group

SUMMARY:
The use of contrast media (CM) poses a risk of post-contrast acute kidney injury (PC-AKI), especially among patients chronic kidney disease (CKD). International guidelines recommend intravenous (IV) hydration with isotonic 0.9% NaCl for three-four hours pre-contrast and four-six hours post-contrast. Recent studies have proven that oral hydration or no hydration is non-inferior to IV hydration in patients with mild to moderate CKD (eGFR 30-60 mL/min/1.73 m2). However, no randomized controlled trials have evaluated alternative hydration methods against the guideline-recommended hydration protocol for the prevention of PC-AKI in high-risk patients with severe CKD (eGFR < 30 mL/min/1.73 m2).

Thus, the main focus of this trial is to evaluate IV hydration vs. oral hydration for their efficacy to prevent of PC-AKI in patients with severe CKD, who are scheduled for an elective contrast-enhanced CT-scan (CECT) with IV contrast-administration.

Our research hypotheses consist of the following:

1. Oral hydration with bottled tap water is non-inferior to IV-hydration with isotonic 0.9% NaCl as renal prophylaxis to prevent PC-AKI in patients with severe CKD referred for an elective IV CECT.
2. NGAL and cfDNA are early and precise plasma and urinary biomarkers of PC-AKI with excellent diagnostic and prognostic accuracy for PC-AKI, dialysis, renal adverse events, hospitalization, progression in CKD-symptoms, and all-cause mortality.

DETAILED DESCRIPTION:
Trial design:

This study is a pragmatic investigator-iniated, single-centre, open-labelled, parallel-group non-inferiority randomized controlled trial with two parallel arms. Patients will randomly be allocated to preventive treatment with IV hydration or oral hydration.

Participants and study setting:

The ENRICH-trial is conducted at Odense University Hospital (OUH), which is a tertiary health-care centre. The referral area covers the region of Southern Denmark, which corresponds to 1.25 million citizens in 22 municipalities of both urban and rural environment. The trial enrols high-risk patients with an eGFR < 30 mL/min/1.73 m2 scheduled for IV CECT using approximately 50-150 mL of CM (GE Healthcare, Omnipaque 500 mL, osmolality 350 mg I/mL).

The study population will consist of patients, who are referred for an elective IV CECT in the work-up for treatment of CVD (e.g., transaortic valve-implantation, ablation, endocarditis etc.) or suspected CVD (e.g., angina etc.), suspected cancer, thoracic/abdominal/urogenital diseases, or cardiovascular work-up before kidney transplantation. Patients referred for an acute or subacute IV CECT with competing etiologies for PC-AKI (e.g., sepsis, acute tubular necrosis, cardiogenic shock etc.) will not be considered eligible for inclusion.

Randomization:

The randomized allocation to preventive treatment with either IV-hydration or oral hydration will be performed in REDCap, which is computer-based tool provided by our collaborator, Open Patient data Explorative Network (OPEN). The randomization sequence list is generated and implemented in the computer-based randomization tool by our data manager and will remain unknown throughout the study period.

The randomization will be performed as 2-4-2 block randomization with stratification for DM-status, CKD-stage (eGFR < 15 mL/min/1.73 m2 or 15-29 mL/min/1.73 m2), and the basis of referral for IV CECT (kidney transplantation or other diseases). Participants are then followed for a 30-day period with standard blood testing for kidney function at two-five days after IV CECT and a 30-day follow-up for the key secondary outcomes.

Definition of PC-AKI:

PC-AKI is defined in accordance with the KDIGO-guidelines, which is a relative increase in serum creatinine (SCr) > 50% from baseline or an absolute increase of SCr > 0.3 mg/dL from baseline.

Course of action:

High-risk patients with severe CKD (eGFR < 30 mL/min/1.73 m2) and a scheduled IV CECT will be considered for eligibility. Eligible patients will be screened according to the study's inclusion/exclusion criteria. Eligibility is assessed from the patient's electronic health record (EHR), which contains data regarding health status and recent test results for evaluation of renal function.

Eligible patients will be presented to the guideline-recommendations for preventive treatment with IV hydration along with blood sampling for evaluation of their renal function < seven days prior to the IV CECT at the time of the scheduling of their IV CECT, according to normal routine at Odense University Hospital. Furthermore, the patients will be presented with a short introduction to this study. If the patient is interested, he/she will be contacted by the lead investigators, after which a verbal consent to participate in the study is obtained (approximately seven to 14 days prior to the scheduled IV CECT).

After the verbal consent is given, the guideline-required evaluation of renal function < seven days prior to their IV CECT will be planned along with an additional blood sample to evaluate the renal function one-three days prior to their IV CECT. Furthermore, blood samples to evaluate renal function will be planned at two-three days, four-five days, and 30 days after IV CECT along with follow-up consultations four-five days and 30 days after IV CECT.

A thorough presentation of the study-information will be given by one of the lead investigators at baseline, while the patient has been informed about the possibility of bringing an assessor of their choice. The information will be delivered in a quiet room, which is solely used to deliver patient information. The lead investigators will make sure that the presentation is given within a reasonable timeframe prior to their scheduled IV CECT.

During the presentation of the study the patient will be informed of the purpose of the study and the written patient information will be sent via e-mail or physically handed to the patient if desired. Patients will be given as much time as wanted to decide if they wish to participate in the study after the oral information has been given. Patients will be offered the possibility to call or physically meet with one of the lead investigators in case of additional questions before signing the informed consent.

Subjects can leave the study at any time for any reason if they wish to do so without any clinical consequences. Signed informed consent will be provided prior to any research procedures. A subject is considered enrolled in the study once the subject is randomized.

Patient data from EHR will be obtained according to the REDCap-database and the study endpoints after the verbal consent is delivered.

Participant retention, follow-up, and withdrawal:

Once a patient is enrolled and randomized, the research group will make every reasonable effort to follow the patient for the entire study period. If the patient fails to attend their appointment for blood sampling to evaluate renal function, the patient will be contacted by telephone, and a new appointment for blood sampling is scheduled within the next 24 hours. The patient will only be excluded from the study after randomization if the patient does not receive the preventive treatment according to the randomization or if the IV CECT is cancelled after randomization and preventive treatment. The rate of loss-to-follow-up for the primary and secondary outcomes are expected to be < 10%.

Variables:

Standard blood parameters to evaluate renal function will be obtained < 90 days, < seven days, one-three days, and at baseline prior to the scheduled IV CECT. Furthermore, an urine sample for albumine/creatinine ratio (mg/g) will be obtained at baseline before CM exposure. The standard blood parameters will also be obtained two-three days and/or four-five days, and 25-40 days after the scheduled IV CECT. Additional blood sampling to evaluate renal function will be performed at seven days and/or 14-21 days after IV CECT if the patient has increasing SCr four-five days after IV CECT consistent with PC-AKI.

The standard blood parameters for patients referred for IV CECT consist of the following: Hemoglobin (mM), erythrocytes (count/L), SCr (μmol/L), eGFR (mL/min/1.73 m2), albumine (μmol/L), sodium (mM), and potassium (mM).

The prospective cohort is followed over a 30-day period for events of dialysis treatment, renal adverse events, hospitalization due to hydration- or contrast-related sequelae (i.e., symptomatic heart failure, arrythmias, renal insufficiency, hyponatremia or hypernatremia), and all-cause mortality.

Progression in CKD-symptoms will be obtained from registration of uremic symptoms through a medical interview at baseline and ≤ 30 days after IV CECT. A trained interviewer will identify any clinical signs of progression in CKD within the 30-day follow-up. Progression in CKD is defined as progression in uremic symptoms, which consist of the following:

- Weight loss, loss of appetite, cramps, nausea, vomiting, pruritus, bruising, fatigue, peripheral edema, impaired consciousness, and changes in sense of taste.

The medical history, medicine use, and echocardiography will be obtained at baseline before initiation of the hydration protocol. The patient will then tend to their IV CECT.

Blood- and urine samples for biomarkers of PC-AKI will be collected before IV CECT and three-four hours after IV CECT.

The admission time is defined as the timespan between the start and the completion of the preventive treatment, which is registered as 'date-month-year-hours-minutes'.

Dates and reasons for hospital admission < 90 days before IV CECT will also be registered along with additional contrast exposure within the 30-day follow-up period after the scheduled IV CECT.

The following parameters will also be obtained for the subgroup of participants, who are referred for a cardiac IV CECT:

* Estimated coronary artery calcification score (CAC-score).
* Stenosis > 50% of the left main coronary artery (LM).
* The grade of stenosis will be analyzed if present in the coronary arteries; LM, left anterior descending artery (LAD), left circumflex artery (LCx), and right coronary artery (RCA).
* Aortic valve calcification (AVC) and mitral annulus calcification (MAC).
* Calcification (Agatson-score) of the aorta (aorta ascendens, arcus aorta, and aorta descendens), the suprarenal and infrarenal aorta, and the renal arteries.
* The diameter of aorta (aorta ascendens, arcus aorta, aorta descendens) and iliac arteries.
* The size of the left atrium (cm2).

Safety:

An interim analysis will be performed after inclusion of 127 patients to evaluate the primary outcomes and the key secondary outcomes. The steering committee will consider terminating the study preliminary if the analyses conclude a significant difference in the incidence of the primary and/or the key secondary outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* eGFR < 30 mL/min/1.73 m2
* Scheduled for elective IV CECT
* Age ≥ 18
* Signed informed consent

Exclusion Criteria:

* Allergy to Iodine
* Pregnancy
* Active dialysis treatment
* Acute infectious or inflammatory disease
* Acute pre- and/or post-renal kidney failure
* Unable to understand study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of PC-AKI | 2-5 days after IV CECT
  The incidence of PC-AKI within the two arms

SECONDARY OUTCOMES:
Incidence of new onset need for dialysis treatment | ≤ 30 days after IV CECT
  The incidence of patients with incident need for dialysis treatment, which is registered from the EHR and/or telephone consultation
Renal adverse events | 25-40 days after IV CECT
  The incidence of renal adverse events defined as a relative increase in SCr > 15% and/or a decrease in eGFR > 15% and/or progression in CKD-stage from CKD-stage IV to CKD-stage Va
Hospitalization due to symptomatic heart failure | ≤ 30 days after IV CECT
  The incidence of patients hospitalized due to symptomatic heart failure, which is registered from the EHR and/or telephone consultation
All-cause mortality | ≤ 30 days after IV CECT
  All-cause mortality, which is registered from the EHR
Hospitalization due to suspected hydration- or contrast-related sequelae | ≤ 30 days after IV CECT
  Hospitalization due to suspected hydration- or contrast-related sequelae (e.g., arrythmias, renal insufficiency, hyponatremia or hypernatremia), which is registered from the EHR and/or telephone consultation
Progression in CKD-symptoms | ≤ 30 days after IV CECT
  Progression in CKD-symptoms within 30 days after IV CECT defined as an increase in number of uremic symptoms compared to number of uremic at baseline within the two arms (see definition of "uremic symptoms" under "Variables" in the detailed description of the trial)
Incidence of PC-AKI based on the criteria from the previously used and most cited definition of PC-AKI | 2-5 days after IV CECT
  The incidence of PC-AKI within the population and the two arms defined as a relative increase in SCr > 25% from baseline or an absolute increase > 0.5 mg/dL
Timepoints of diagnosis for PC-AKI | 2-5 days after IV CECT
  The difference in PC-AKI diagnosed two-three days after IV CECT and four-five days after IV CECT within the population and the two arms
Number of patients with normalization of PC-AKI | ≤ 40 days after IV CECT
  Number of participants with normalization of PC-AKI within study population and the two arms defined as a decline in SCr below the criteria for PC-AKI
Mean changes in SCr | SCr is measured on the following time-points (days from baseline): -89 to -seven days, -six to -four days, -three to -one days, 0 days (baseline), +two to three days, +four to five days, and +25 to +40 days
  Mean changes in SCr from baseline at different timepoints within the study population and the two arms
Mean changes in eGFR. | eGFR is measured on the following time-points (days from baseline): -89 to -seven days, -six to -four days, -three to -one days, 0 days (baseline), +two to three days, +four to five days, and +25 to +40 days
  Mean changes in eGFR from baseline at different timepoints within the study population and the two arms
The effect of hydration on standard blood parameters | Standard blood parameters will be obtained after IV CECT at +two to three days and/or +four to five days, and +25 to +40 days from baseline
  Mean changes in standard blood parameters within the two arms. Standard blood parameters are the following: Hemoglobin (mM), erythrocytes (count/L), SCr (micromole/L), eGFR (mL/min/1.73 m2), albumine (micromole/L), sodium (mM), and potassium (mM)
Mean values of plasma and urinary NGAL and cell-free DNA | In-hospital: Before initiation of the hydration protocol and the IV CECT (baseline) and 4 hours after IV CECT
  Mean values of plasma and urinary NGAL (μg/mg) and cell-free DNA (ng/mg) at baseline and 4 hours after IV CECT
Mean changes of plasma and urinary NGAL and cell-free DNA | In-hospital: Before initiation of the hydration protocol and the IV CECT (baseline) and 4 hours after IV CECT
  Mean changes in plasma and urinary NGAL (μg/mg) and cell-free DNA (ng/mg) from baseline (0 hours) to four hours after IV CECT
The diagnostic and prognostic accuracy of plasma and urinary NGAL and cell-free DNA | In-hospital: Before initiation of the hydration protocol and the IV CECT (baseline) and 4 hours after IV CECT
  Sensitivities, specificities, negative predictive values, positive predictive values, negative likelihood-ratios, and positive likelihood-ratios of plasma and urinary NGAL (μg/mg) and cell-free DNA (ng/mg) based on the most optimal cut-off point for each biomarker based on Receiver Operating Characteristics-Curves (ROC-curves) and their corresponding Area Under Curve (AUC). The most optimal cut-off is defined as the closest point on the ROC-curves, at which the sensitivity = specificity = 1.0
The diagnostic and prognostic accuracy of plasma and urinary NGAL and cell-free DNA | In-hospital: Before initiation of the hydration protocol and the IV CECT (baseline) and 4 hours after IV CECT
  Assesment of the most optimal cut-off point for each biomarker based on Receiver Operating Characteristics-Curves (ROC-curves) and their corresponding Area Under Curve (AUC). The most optimal cut-off is defined as the closest point on the ROC-curves, at which the sensitivity = specificity = 1.0
The diagnostic and prognostic accuracy of plasma and urinary NGAL and cell-free DNA | In-hospital: Before initiation of the hydration protocol and the IV CECT (baseline) and 4 hours after IV CECT
  The correlation between SCr and plasma and urinary NGAL (μg/mg) and cell-free DNA (ng/mg) will be illustrated in Scatter Plots.
Cost-effectiveness | 1 day (at the day of the patient's scheduled cardiac CT)
  The use of resources (presented in DKK, EUR, and USD) for IV-hydration and oral hydration within the two arms are calculated from the following parameters: The cost of occupying a hospital bed per hour (nursing, staff salaries etc.), IV-drip, and hydration bags with saline or bottled tap water.
Time-effectiveness of the two hydration protocols. | In-hospital: Starting 1-3 hours before IV CECT and lasting maximally until 4 hours after IV CECT
  The two hydration methods are compared for the amount of time (hours and minutes) from initiation to completion hydration protocols.
Risk of PC-AKI according to the size of the kidneys | 2-5 days after IV CECT
  The size of the right and left kidney will be measured and indexed to the body-size of the patient and analyzed as a risk factor for the occurence of PC-AKI

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Odense C, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available in an anonymous format in accordance with the legislations from GDPR upon reasonable request.
  Rules for external researchers to apply for and access data will be laid out towards the end of the study.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: TBA
Access Criteria: TBA

REFERENCES:
- [Background] Christiansen C. X-ray contrast media--an overview. Toxicology. 2005 Apr 15;209(2):185-7. doi: 10.1016/j.tox.2004.12.020. PMID 15767033
- [Background] van der Molen AJ, Reimer P, Dekkers IA, Bongartz G, Bellin MF, Bertolotto M, Clement O, Heinz-Peer G, Stacul F, Webb JAW, Thomsen HS. Post-contrast acute kidney injury - Part 1: Definition, clinical features, incidence, role of contrast medium and risk factors : Recommendations for updated ESUR Contrast Medium Safety Committee guidelines. Eur Radiol. 2018 Jul;28(7):2845-2855. doi: 10.1007/s00330-017-5246-5. Epub 2018 Feb 9. PMID 29426991
- [Background] van der Molen AJ, Reimer P, Dekkers IA, Bongartz G, Bellin MF, Bertolotto M, Clement O, Heinz-Peer G, Stacul F, Webb JAW, Thomsen HS. Post-contrast acute kidney injury. Part 2: risk stratification, role of hydration and other prophylactic measures, patients taking metformin and chronic dialysis patients : Recommendations for updated ESUR Contrast Medium Safety Committee guidelines. Eur Radiol. 2018 Jul;28(7):2856-2869. doi: 10.1007/s00330-017-5247-4. Epub 2018 Feb 7. PMID 29417249
- [Background] McCullough PA, Choi JP, Feghali GA, Schussler JM, Stoler RM, Vallabahn RC, Mehta A. Contrast-Induced Acute Kidney Injury. J Am Coll Cardiol. 2016 Sep 27;68(13):1465-1473. doi: 10.1016/j.jacc.2016.05.099. PMID 27659469
- [Background] Mehran R, Nikolsky E. Contrast-induced nephropathy: definition, epidemiology, and patients at risk. Kidney Int Suppl. 2006 Apr;(100):S11-5. doi: 10.1038/sj.ki.5000368. PMID 16612394
- [Background] Mehran R, Dangas GD, Weisbord SD. Contrast-Associated Acute Kidney Injury. N Engl J Med. 2019 May 30;380(22):2146-2155. doi: 10.1056/NEJMra1805256. No abstract available. PMID 31141635
- [Background] Davenport MS, Perazella MA, Yee J, Dillman JR, Fine D, McDonald RJ, Rodby RA, Wang CL, Weinreb JC. Use of Intravenous Iodinated Contrast Media in Patients with Kidney Disease: Consensus Statements from the American College of Radiology and the National Kidney Foundation. Radiology. 2020 Mar;294(3):660-668. doi: 10.1148/radiol.2019192094. Epub 2020 Jan 21. PMID 31961246
- [Background] McCullough PA, Adam A, Becker CR, Davidson C, Lameire N, Stacul F, Tumlin J; CIN Consensus Working Panel. Risk prediction of contrast-induced nephropathy. Am J Cardiol. 2006 Sep 18;98(6A):27K-36K. doi: 10.1016/j.amjcard.2006.01.022. Epub 2006 Feb 23. PMID 16949378
- [Background] Jha V, Garcia-Garcia G, Iseki K, Li Z, Naicker S, Plattner B, Saran R, Wang AY, Yang CW. Chronic kidney disease: global dimension and perspectives. Lancet. 2013 Jul 20;382(9888):260-72. doi: 10.1016/S0140-6736(13)60687-X. Epub 2013 May 31. PMID 23727169
- [Background] Nash K, Hafeez A, Hou S. Hospital-acquired renal insufficiency. Am J Kidney Dis. 2002 May;39(5):930-6. doi: 10.1053/ajkd.2002.32766. PMID 11979336
- [Background] Rihal CS, Textor SC, Grill DE, Berger PB, Ting HH, Best PJ, Singh M, Bell MR, Barsness GW, Mathew V, Garratt KN, Holmes DR Jr. Incidence and prognostic importance of acute renal failure after percutaneous coronary intervention. Circulation. 2002 May 14;105(19):2259-64. doi: 10.1161/01.cir.0000016043.87291.33. PMID 12010907
- [Background] Chertow GM, Burdick E, Honour M, Bonventre JV, Bates DW. Acute kidney injury, mortality, length of stay, and costs in hospitalized patients. J Am Soc Nephrol. 2005 Nov;16(11):3365-70. doi: 10.1681/ASN.2004090740. Epub 2005 Sep 21. PMID 16177006
- [Background] Katzberg RW, Newhouse JH. Intravenous contrast medium-induced nephrotoxicity: is the medical risk really as great as we have come to believe? Radiology. 2010 Jul;256(1):21-8. doi: 10.1148/radiol.10092000. No abstract available. PMID 20574082
- [Background] Solomon R. Contrast-induced acute kidney injury: is there a risk after intravenous contrast? Clin J Am Soc Nephrol. 2008 Sep;3(5):1242-3. doi: 10.2215/CJN.03470708. Epub 2008 Aug 13. No abstract available. PMID 18701610
- [Background] Ellis JH, Cohan RH. Reducing the risk of contrast-induced nephropathy: a perspective on the controversies. AJR Am J Roentgenol. 2009 Jun;192(6):1544-9. doi: 10.2214/AJR.09.2368. PMID 19457817
- [Background] Rao QA, Newhouse JH. Risk of nephropathy after intravenous administration of contrast material: a critical literature analysis. Radiology. 2006 May;239(2):392-7. doi: 10.1148/radiol.2392050413. Epub 2006 Mar 16. PMID 16543592
- [Background] McDonald JS, McDonald RJ, Carter RE, Katzberg RW, Kallmes DF, Williamson EE. Risk of intravenous contrast material-mediated acute kidney injury: a propensity score-matched study stratified by baseline-estimated glomerular filtration rate. Radiology. 2014 Apr;271(1):65-73. doi: 10.1148/radiol.13130775. Epub 2014 Jan 16. PMID 24475854
- [Background] McDonald JS, McDonald RJ, Lieske JC, Carter RE, Katzberg RW, Williamson EE, Kallmes DF. Risk of Acute Kidney Injury, Dialysis, and Mortality in Patients With Chronic Kidney Disease After Intravenous Contrast Material Exposure. Mayo Clin Proc. 2015 Aug;90(8):1046-53. doi: 10.1016/j.mayocp.2015.05.016. PMID 26250726
- [Background] James MT, Samuel SM, Manning MA, Tonelli M, Ghali WA, Faris P, Knudtson ML, Pannu N, Hemmelgarn BR. Contrast-induced acute kidney injury and risk of adverse clinical outcomes after coronary angiography: a systematic review and meta-analysis. Circ Cardiovasc Interv. 2013 Feb;6(1):37-43. doi: 10.1161/CIRCINTERVENTIONS.112.974493. Epub 2013 Jan 15. PMID 23322741
- [Background] Davenport MS, Khalatbari S, Dillman JR, Cohan RH, Caoili EM, Ellis JH. Contrast material-induced nephrotoxicity and intravenous low-osmolality iodinated contrast material. Radiology. 2013 Apr;267(1):94-105. doi: 10.1148/radiol.12121394. Epub 2013 Jan 29. PMID 23360737
- [Background] McDonald JS, McDonald RJ, Comin J, Williamson EE, Katzberg RW, Murad MH, Kallmes DF. Frequency of acute kidney injury following intravenous contrast medium administration: a systematic review and meta-analysis. Radiology. 2013 Apr;267(1):119-28. doi: 10.1148/radiol.12121460. Epub 2013 Jan 14. PMID 23319662
- [Background] McDonald RJ, McDonald JS, Bida JP, Carter RE, Fleming CJ, Misra S, Williamson EE, Kallmes DF. Intravenous contrast material-induced nephropathy: causal or coincident phenomenon? Radiology. 2013 Apr;267(1):106-18. doi: 10.1148/radiol.12121823. Epub 2013 Jan 29. PMID 23360742
- [Background] McDonald RJ, McDonald JS, Carter RE, Hartman RP, Katzberg RW, Kallmes DF, Williamson EE. Intravenous contrast material exposure is not an independent risk factor for dialysis or mortality. Radiology. 2014 Dec;273(3):714-25. doi: 10.1148/radiol.14132418. Epub 2014 Sep 9. PMID 25203000
- [Background] Nijssen EC, Nelemans PJ, Rennenberg RJ, van Ommen V, Wildberger JE. Evaluation of Safety Guidelines on the Use of Iodinated Contrast Material: Conundrum Continued. Invest Radiol. 2018 Oct;53(10):616-622. doi: 10.1097/RLI.0000000000000479. PMID 29762257
- [Background] Geenen RW, Kingma HJ, van der Molen AJ. Contrast-induced nephropathy: pharmacology, pathophysiology and prevention. Insights Imaging. 2013 Dec;4(6):811-20. doi: 10.1007/s13244-013-0291-3. Epub 2013 Oct 3. PMID 24092564
- [Background] Newhouse JH, Kho D, Rao QA, Starren J. Frequency of serum creatinine changes in the absence of iodinated contrast material: implications for studies of contrast nephrotoxicity. AJR Am J Roentgenol. 2008 Aug;191(2):376-82. doi: 10.2214/AJR.07.3280. PMID 18647905
- [Background] Waikar SS, Bonventre JV. Creatinine kinetics and the definition of acute kidney injury. J Am Soc Nephrol. 2009 Mar;20(3):672-9. doi: 10.1681/ASN.2008070669. Epub 2009 Feb 25. PMID 19244578
- [Background] Seibert FS, Heringhaus A, Pagonas N, Rudolf H, Rohn B, Bauer F, Timmesfeld N, Trappe HJ, Babel N, Westhoff TH. Biomarkers in the prediction of contrast media induced nephropathy - the BITCOIN study. PLoS One. 2020 Jul 16;15(7):e0234921. doi: 10.1371/journal.pone.0234921. eCollection 2020. PMID 32673348
- [Background] Filiopoulos V, Biblaki D, Vlassopoulos D. Neutrophil gelatinase-associated lipocalin (NGAL): a promising biomarker of contrast-induced nephropathy after computed tomography. Ren Fail. 2014 Jul;36(6):979-86. doi: 10.3109/0886022X.2014.900429. Epub 2014 Mar 27. PMID 24673459
- [Background] Lacquaniti A, Buemi F, Lupica R, Giardina C, Mure G, Arena A, Visalli C, Baldari S, Aloisi C, Buemi M. Can neutrophil gelatinase-associated lipocalin help depict early contrast material-induced nephropathy? Radiology. 2013 Apr;267(1):86-93. doi: 10.1148/radiol.12120578. Epub 2013 Jan 7. PMID 23297321
- [Background] Quintavalle C, Anselmi CV, De Micco F, Roscigno G, Visconti G, Golia B, Focaccio A, Ricciardelli B, Perna E, Papa L, Donnarumma E, Condorelli G, Briguori C. Neutrophil Gelatinase-Associated Lipocalin and Contrast-Induced Acute Kidney Injury. Circ Cardiovasc Interv. 2015 Sep;8(9):e002673. doi: 10.1161/CIRCINTERVENTIONS.115.002673. PMID 26333343
- [Background] Nickolas TL, Schmidt-Ott KM, Canetta P, Forster C, Singer E, Sise M, Elger A, Maarouf O, Sola-Del Valle DA, O'Rourke M, Sherman E, Lee P, Geara A, Imus P, Guddati A, Polland A, Rahman W, Elitok S, Malik N, Giglio J, El-Sayegh S, Devarajan P, Hebbar S, Saggi SJ, Hahn B, Kettritz R, Luft FC, Barasch J. Diagnostic and prognostic stratification in the emergency department using urinary biomarkers of nephron damage: a multicenter prospective cohort study. J Am Coll Cardiol. 2012 Jan 17;59(3):246-55. doi: 10.1016/j.jacc.2011.10.854. PMID 22240130
- [Background] Liu C, Debnath N, Mosoyan G, Chauhan K, Vasquez-Rios G, Soudant C, Menez S, Parikh CR, Coca SG. Systematic Review and Meta-Analysis of Plasma and Urine Biomarkers for CKD Outcomes. J Am Soc Nephrol. 2022 Sep;33(9):1657-1672. doi: 10.1681/ASN.2022010098. Epub 2022 Jul 20. PMID 35858701
- [Background] Haase M, Bellomo R, Devarajan P, Schlattmann P, Haase-Fielitz A; NGAL Meta-analysis Investigator Group. Accuracy of neutrophil gelatinase-associated lipocalin (NGAL) in diagnosis and prognosis in acute kidney injury: a systematic review and meta-analysis. Am J Kidney Dis. 2009 Dec;54(6):1012-24. doi: 10.1053/j.ajkd.2009.07.020. Epub 2009 Oct 21. PMID 19850388
- [Background] Merkle J, Daka A, Deppe AC, Wahlers T, Paunel-Gorgulu A. High levels of cell-free DNA accurately predict late acute kidney injury in patients after cardiac surgery. PLoS One. 2019 Jun 18;14(6):e0218548. doi: 10.1371/journal.pone.0218548. eCollection 2019. PMID 31211810
- [Background] Celec P, Vlkova B, Laukova L, Babickova J, Boor P. Cell-free DNA: the role in pathophysiology and as a biomarker in kidney diseases. Expert Rev Mol Med. 2018 Jan 18;20:e1. doi: 10.1017/erm.2017.12. PMID 29343314
- [Background] Sun SQ, Zhang T, Ding D, Zhang WF, Wang XL, Sun Z, Hu LH, Qin SY, Shen LH, He B. Circulating MicroRNA-188, -30a, and -30e as Early Biomarkers for Contrast-Induced Acute Kidney Injury. J Am Heart Assoc. 2016 Aug 15;5(8):e004138. doi: 10.1161/JAHA.116.004138. PMID 27528406
- [Background] Homolova J, Janovicova L, Konecna B, Vlkova B, Celec P, Tothova L, Babickova J. Plasma Concentrations of Extracellular DNA in Acute Kidney Injury. Diagnostics (Basel). 2020 Mar 11;10(3):152. doi: 10.3390/diagnostics10030152. PMID 32168933
- [Background] Jancuska A, Potocarova A, Kovalcikova AG, Podracka L, Babickova J, Celec P, Tothova L. Dynamics of Plasma and Urinary Extracellular DNA in Acute Kidney Injury. Int J Mol Sci. 2022 Mar 21;23(6):3402. doi: 10.3390/ijms23063402. PMID 35328821
- [Background] Coimbra S, Rocha S, Nascimento H, Valente MJ, Catarino C, Rocha-Pereira P, Sameiro-Faria M, Oliveira JG, Madureira J, Fernandes JC, Miranda V, Belo L, Bronze-da-Rocha E, Santos-Silva A. Cell-free DNA as a marker for the outcome of end-stage renal disease patients on haemodialysis. Clin Kidney J. 2020 Aug 24;14(5):1371-1378. doi: 10.1093/ckj/sfaa115. eCollection 2021 May. PMID 33959266
- [Background] Nijssen EC, Rennenberg RJ, Nelemans PJ, Essers BA, Janssen MM, Vermeeren MA, Ommen VV, Wildberger JE. Prophylactic hydration to protect renal function from intravascular iodinated contrast material in patients at high risk of contrast-induced nephropathy (AMACING): a prospective, randomised, phase 3, controlled, open-label, non-inferiority trial. Lancet. 2017 Apr 1;389(10076):1312-1322. doi: 10.1016/S0140-6736(17)30057-0. Epub 2017 Feb 21. PMID 28233565
- [Background] Sebastia C, Paez-Carpio A, Guillen E, Pano B, Garcia-Cinca D, Poch E, Oleaga L, Nicolau C. Oral hydration compared to intravenous hydration in the prevention of post-contrast acute kidney injury in patients with chronic kidney disease stage IIIb: A phase III non-inferiority study (NICIR study). Eur J Radiol. 2021 Mar;136:109509. doi: 10.1016/j.ejrad.2020.109509. Epub 2021 Jan 14. PMID 33516141
- [Background] Agarwal SK, Mohareb S, Patel A, Yacoub R, DiNicolantonio JJ, Konstantinidis I, Pathak A, Fnu S, Annapureddy N, Simoes PK, Kamat S, El-Hayek G, Prasad R, Kumbala D, Nascimento RM, Reilly JP, Nadkarni GN, Benjo AM. Systematic oral hydration with water is similar to parenteral hydration for prevention of contrast-induced nephropathy: an updated meta-analysis of randomised clinical data. Open Heart. 2015 Oct 5;2(1):e000317. doi: 10.1136/openhrt-2015-000317. eCollection 2015. PMID 26468404
- [Background] Cheungpasitporn W, Thongprayoon C, Brabec BA, Edmonds PJ, O'Corragain OA, Erickson SB. Oral hydration for prevention of contrast-induced acute kidney injury in elective radiological procedures: a systematic review and meta-analysis of randomized controlled trials. N Am J Med Sci. 2014 Dec;6(12):618-24. doi: 10.4103/1947-2714.147977. PMID 25599049
- [Background] Dong M, Jiao Z, Liu T, Guo F, Li G. Effect of administration route on the renal safety of contrast agents: a meta-analysis of randomized controlled trials. J Nephrol. 2012 May-Jun;25(3):290-301. doi: 10.5301/jn.5000067. PMID 22252847
- [Background] Hiremath S, Akbari A, Shabana W, Fergusson DA, Knoll GA. Prevention of contrast-induced acute kidney injury: is simple oral hydration similar to intravenous? A systematic review of the evidence. PLoS One. 2013;8(3):e60009. doi: 10.1371/journal.pone.0060009. Epub 2013 Mar 26. PMID 23555863
- [Background] Timal RJ, Kooiman J, Sijpkens YWJ, de Vries JPM, Verberk-Jonkers IJAM, Brulez HFH, van Buren M, van der Molen AJ, Cannegieter SC, Putter H, van den Hout WB, Jukema JW, Rabelink TJ, Huisman MV. Effect of No Prehydration vs Sodium Bicarbonate Prehydration Prior to Contrast-Enhanced Computed Tomography in the Prevention of Postcontrast Acute Kidney Injury in Adults With Chronic Kidney Disease: The Kompas Randomized Clinical Trial. JAMA Intern Med. 2020 Apr 1;180(4):533-541. doi: 10.1001/jamainternmed.2019.7428. PMID 32065601
- [Background] Yoshikawa D, Isobe S, Sato K, Ohashi T, Fujiwara Y, Ohyama H, Ishii H, Murohara T. Importance of oral fluid intake after coronary computed tomography angiography: an observational study. Eur J Radiol. 2011 Jan;77(1):118-22. doi: 10.1016/j.ejrad.2009.07.011. Epub 2009 Aug 19. PMID 19695806
- [Background] Aycock RD, Westafer LM, Boxen JL, Majlesi N, Schoenfeld EM, Bannuru RR. Acute Kidney Injury After Computed Tomography: A Meta-analysis. Ann Emerg Med. 2018 Jan;71(1):44-53.e4. doi: 10.1016/j.annemergmed.2017.06.041. Epub 2017 Aug 12. PMID 28811122
- [Background] Kim SM, Cha RH, Lee JP, Kim DK, Oh KH, Joo KW, Lim CS, Kim S, Kim YS. Incidence and outcomes of contrast-induced nephropathy after computed tomography in patients with CKD: a quality improvement report. Am J Kidney Dis. 2010 Jun;55(6):1018-25. doi: 10.1053/j.ajkd.2009.10.057. Epub 2010 Jan 25. PMID 20097462
- [Background] Wu MJ, Tsai SF. Patients with Different Stages of Chronic Kidney Disease Undergoing Intravenous Contrast-Enhanced Computed Tomography-The Incidence of Contrast-Associated Acute Kidney Injury. Diagnostics (Basel). 2022 Mar 30;12(4):864. doi: 10.3390/diagnostics12040864. PMID 35453910
- [Background] LaBounty TM, Shah M, Raman SV, Lin FY, Berman DS, Min JK. Within-hospital and 30-day outcomes in 107,994 patients undergoing invasive coronary angiography with different low-osmolar iodinated contrast media. Am J Cardiol. 2012 Jun 1;109(11):1594-9. doi: 10.1016/j.amjcard.2012.01.380. Epub 2012 Mar 20. PMID 22440116
- [Background] Kift RL, Messenger MP, Wind TC, Hepburn S, Wilson M, Thompson D, Smith MW, Sturgeon C, Lewington AJ, Selby PJ, Banks RE. A comparison of the analytical performance of five commercially available assays for neutrophil gelatinase-associated lipocalin using urine. Ann Clin Biochem. 2013 May;50(Pt 3):236-44. doi: 10.1258/acb.2012.012117. PMID 23605129
- [Background] Magnusson NE, Hornum M, Jorgensen KA, Hansen JM, Bistrup C, Feldt-Rasmussen B, Flyvbjerg A. Plasma neutrophil gelatinase associated lipocalin (NGAL) is associated with kidney function in uraemic patients before and after kidney transplantation. BMC Nephrol. 2012 Feb 10;13:8. doi: 10.1186/1471-2369-13-8. PMID 22325322
- [Background] McCullough PA. Contrast-induced acute kidney injury. J Am Coll Cardiol. 2008 Apr 15;51(15):1419-28. doi: 10.1016/j.jacc.2007.12.035. PMID 18402894
- [Background] Zhang W, Zhang J, Yang B, Wu K, Lin H, Wang Y, Zhou L, Wang H, Zeng C, Chen X, Wang Z, Zhu J, Songming C. Effectiveness of oral hydration in preventing contrast-induced acute kidney injury in patients undergoing coronary angiography or intervention: a pairwise and network meta-analysis. Coron Artery Dis. 2018 Jun;29(4):286-293. doi: 10.1097/MCA.0000000000000607. PMID 29381498
- [Background] Dussol B, Morange S, Loundoun A, Auquier P, Berland Y. A randomized trial of saline hydration to prevent contrast nephropathy in chronic renal failure patients. Nephrol Dial Transplant. 2006 Aug;21(8):2120-6. doi: 10.1093/ndt/gfl133. Epub 2006 Apr 12. PMID 16611682
- [Background] Martin-Moreno PL, Varo N, Martinez-Anso E, Martin-Calvo N, Sayon-Orea C, Bilbao JI, Garcia-Fernandez N. Comparison of Intravenous and Oral Hydration in the Prevention of Contrast-Induced Acute Kidney Injury in Low-Risk Patients: A Randomized Trial. Nephron. 2015;131(1):51-8. doi: 10.1159/000438907. Epub 2015 Aug 26. PMID 26336919
- [Background] Faggioni M, Mehran R. Preventing Contrast-induced Renal Failure: A Guide. Interv Cardiol. 2016 Oct;11(2):98-104. doi: 10.15420/icr.2016:10:2. PMID 29588714
- [Derived] Ravn EJ, Hasific S, Thomassen M, Hjortebjerg R, Bach Laursen K, Diederichsen A, Bistrup C, Ovrehus KA. Intravenous versus oral hydration to reduce the risk of postcontrast acute kidney injury after intravenous contrast-enhanced CT in patients with severe chronic kidney disease (ENRICH): a study protocol for a single-centre, parallel-group, open-labelled non-inferiority randomised controlled trial in Denmark. BMJ Open. 2023 Sep 12;13(9):e074057. doi: 10.1136/bmjopen-2023-074057. PMID 37699636
- See also: OECD (2022), Computed tomography (CT) exams (indicator). doi: 10.1787/3c994537-en (Accessed on 02 February 2022). — https://data.oecd.org/healthcare/computed-tomography-ct-exams.htm
- See also: Kidney Disease Improving Global Outcomes. KDIGO clinical practice guideline for acute kidney injury — http://kdigo.org/home/guidelines/
- See also: European Society of Urogenital Radiology's Guidelines on Contrast Agents. — https://www.esur.org/fileadmin/content/2019/ESUR_Guidelines_10.0_Final_Version.pdf
- See also: American College of Radiology - Manual on Contrast Media 2023 — https://www.acr.org/-/media/acr/files/clinical-resources/contrast_media.pdf